CLINICAL TRIAL: NCT04869605
Title: 1,5 Anhydroglucitol and 1,5 Anhydroglucitol / Glycated Hemoglobin Ratio as a Potential Biomarker for Islet β-cell Function and Insulin Resistance Among Patients With Type 2 Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mona Youssry Helmy, Lecturer of internal medicine, Cairo University
Other Study IDs: N-26-2021
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 1,5 Anhydroglucitol and 1,5 Anhydroglucitol / Glycated Hemoglobin ratio — the role of 1,5 anhydroglucitol and 1,5 anhydroglucitol / HbA1c ratio as a potential biomarker for islet β-cell function and insulin resistance among patients with type 2 diabetes

SUMMARY:
Hyperglycemia is a major risk factor for the micro- and macro-vascular complications of diabetes . Lowering blood glucose levels has been shown to reduce the incidence of diabetes complications.

Therefore, there is a need for a simple surrogate biochemical marker for glycemic variability. Glycated hemoglobin (HbA1c) is the standard clinical measurement used to monitor glycemic status and is recommended to assess control of diabetes over the preceding 2-3 months. However, being a measure of mean glucose, it does not reflect glucose variability.

It is well known that insulin secretion defects of islet β cells and/or tissue insensitivity to insulin are common pathophysiological mechanisms of diabetes mellitus (DM) .

The elevation in the blood glucose level usually represents the degree of glucose metabolism disorder, which is generally assessed by glycated hemoglobin A1c ( HbA1c) and indirectly reflects the extent of β-cell function damage .

In the recent years, 1,5-anhydroglucitol (1,5-AG) has received attention as a short-term blood glucose index that reflects the average blood glucose level 1,5 AG reflects the average maximum blood glucose level during the past 1-2 weeks and is reported to be a more sensitive marker of glucose variability and postprandial hyperglycemia than HbA1c, even for patients with prediabetes and for those with well or moderately controlled diabetes .

(1,5 AG ) is structurally similar to glucose . Due to this similarity, glucose inhibits renal reabsorption of 1,5 AG by competitive inhibition ,resulting in an inverse correlation of 1,5 AG with hyperglycemia .

1,5-AG levels are acting as an effective supplement to HbA1c. Additionally, previous study showed that 1,5-AG and HbA1c had opposite curves with increasing blood glucose levels; specifically, with the increase in HbA1c levels, 1,5-AG levels decreased significantly . Therefore, we speculate a ratio of 1,5- AG / HB A1C in relation to islet β-cell function and insulin resistance.

The aim of our study was to evaluate the role of 1,5 anhydroglucitol and 1,5 anhydroglucitol / HbA1c ratio as a potential biomarker for islet β-cell function and insulin resistance among patients with type 2 diabetes .

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 20 to 70 years old with controlled and uncontrolled type 2 DM.

Exclusion Criteria:

* : type 1 DM,
* thyroid dysfunction,
* chronic kidney disease,
* chronic liver disease,
* cancer patients,
* cystic fibrosis,
* acute and chronic infection and
* pregnancy

Ages: 20 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A case control study including 90 subjects aged 20 to 70 years, 45 healthy subjects as a control group and 45 patients with type 2 DM .Patients will be collected from the endocrinology outpatient clinic, Kasr El Ainy, Cairo University. Patients will be divided into 2 groups, (group I) 45 patients with type 2 DM and (group II) 45 non DM as control group.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
the role of 1,5 anhydroglucitol and 1,5 anhydroglucitol / HbA1c ratio as a potential biomarker for islet β-cell function and insulin resistance among patients with type 2 diabetes | 6 months
  1,5 anhydroglucitol serum level, V level and 1,5 anhydroglucitol / HbA1c ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: No
not to share

REFERENCES:
- [Background] -Janssen J, van den Berg E, Zinman B , Espeland MA , Geijselaers S LC et al., (2019) . HbA(1c), insulin resistance, and β-cell function in relation to cognitive function in type 2 diabetes: the CAROLINA Cognition Substudy. Diabetes Care 42(1):e1-e3. -Kanat M, Winnier D, Norton L, Arar N, Jenkinson C, Defronzo RA et al ., (2011) . The relationship between {beta}-cell function and glycated hemoglobin: results from the veterans administration genetic epidemiology study. Diabetes Care. 2011 Apr;34(4):1006-10. -Kim MJ, Jung HS, Hwang-Bo Y, Cho SW, Jang HC, Kim SY et al ., (2013) . Evaluation of 1,5-anhydroglucitol as a marker for glycemic variability in patients with type 2 diabetes mellitus. Acta Diabetol. 2013;50:505-10.